CLINICAL TRIAL: NCT06020001
Title: Clinical Evaluation of the AP203 Plant Extract Mixture in Adult Patients With Increased Incidence of Viral and/or Bacterial Upper Respiratory Tract Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AronPharma Sp. z o. o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 06-AP-COV
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Upper Respiratory Tract Infection Bacterial
Keywords: Upper Respiratory Tract Infections; Bacterial Infections; Viral Infections; RESCOVIN; Plant extract; Chokeberry extract; Echinacea extract
MeSH Terms: conditions — Respiratory Tract Infections; Bacterial Infections; Virus Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AP203 mixture (RESCOVIN®) in capsule form (Experimental): Patients with an increased incidence of upper respiratory tract infection
  Interventions: Dietary Supplement: AP203 mixture (RESCOVIN®)
- AP203 mixture (RESCOVIN®) in syrup form (Experimental): Patients with an increased incidence of upper respiratory tract infection
  Interventions: Dietary Supplement: AP203 mixture (RESCOVIN®)
- Placebo (Placebo Comparator): Patients with an increased incidence of upper respiratory tract infection
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: AP203 mixture (RESCOVIN®) — Polyphenol-rich plant extracts Twice a day
  Arms: AP203 mixture (RESCOVIN®) in capsule form
Dietary Supplement: AP203 mixture (RESCOVIN®) — Polyphenol-rich plant extracts Twice a day
  Arms: AP203 mixture (RESCOVIN®) in syrup form
Other: Placebo — Twice a day
  Arms: Placebo

SUMMARY:
The aim of the study was to assess the efficacy and safety of AP203 preparation (RESCOVIN®) in a group of patients with increased incidence to viral and/or bacterial upper respiratory tract infections.

DETAILED DESCRIPTION:
Randomized, double-blind, cross over study conducted under medical supervision on 1) group of 30 patients receiving AP203 mixture in capsule form and 2) group of 30 receiving placebo. After a washout period a group receiving placebo receiver AP203 mixture in syrup form.

The study group was adult patients with an increased incidence of upper respiratory tract infection. During the study, the effect of a mixture of AP203 extracts (RESCOVIN®) on markers of inflammation and oxidative stress and the effect on the incidence of upper respiratory tract infections was assessed.

ELIGIBILITY:
Inclusion Criteria:

* Women and men, 18-70 years old
* Healthy patients at the time of enrollment to the study (without active upper respiratory tract infection)
* Presence of 2 or more episodes of upper respiratory tract infections or >=2 episodes of cold during the year
* Patients with chronic upper respiratory tract diseases including bronchial asthma
* Signed informed consent
* Women: contraception or postmenopausal age

Exclusion Criteria:

* Intake of supplements containing plant extracts, polyphenols or anthocyanins for the 3 months prior to the study initiation
* Acute inflammation
* Oral immunosuppressive drugs
* Steroid, anti-allergic drugs in exacerbations of chronic disease at least 2 months from the start of study participation
* Antibiotic therapy 1 month prior to study initiation
* Participation in another clinical trial;
* Oncological disease, autoimmune disease, severe liver dysfunction, tuberculosis, leukaemia, multiple sclerosis, AIDS, rheumatoid arthritis, organ transplantation;
* Hypersensitivity/allergy to any of the ingredients of the product, allergy to plants of the Asteraceae family (e.g. chamomile, calendula);
* Women who are pregnant or planning to become pregnant during the study period;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Efficacy and safety of AP203 | Baseline, 2 months, 4 months, 6 months
  Clinical evaluation of the efficacy and safety of AP203, in a group of patients with an increased incidence of viral and/or bacterial upper respiratory tract infections.

SECONDARY OUTCOMES:
hsCRP level | Baseline, 2 months, 4 months, 6 months
  Comparison of hsCRP level
8-iso-PGF2IsoP level | Baseline, 2 months, 4 months, 6 months
  Comparison of 8-iso-PGF2IsoP level
Cold Intensity Score | Baseline, 2 months, 4 months, 6 months
  Comparison of Cold Intensity Score (CIS) values

CONTACTS AND LOCATIONS:
Locations (1):
- Pomorskie Centrum Reumatologiczne im. dr Jadwigi Titz-Kosko, Sopot, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zima K, Sochocka M, Ochnik M, Khaidakov B, Lemke K, Kowalczyk P. Therapeutic Potential of a Natural Blend of Aronia melancarpa, Lonicera caerulea, and Echinacea purpurea Extracts in Treating Upper Respiratory Tract Infections: Preliminary Clinical and In Vitro Immunomodulatory Insights. Int J Mol Sci. 2024 Dec 15;25(24):13436. doi: 10.3390/ijms252413436. PMID 39769201